CLINICAL TRIAL: NCT06045936
Title: Sciatic Block in Contralateral Limb for Treatment of Refractory Phantom and Residual Limb Pain; a Double-Blind Randomized Controlled Trial
Brief Title: A Study of Contralateral Limb Block
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Cole W. Cheney, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-010792
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Limb Pain, Phantom
MeSH Terms: conditions — Phantom Limb | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine Group (Experimental): Subjects will receive a lidocaine injection in the back of their residual limb.
  Interventions: Drug: Lidocaine
- Sham Group (Placebo Comparator): Subjects will receive a placebo injection in the back of their residual limb.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — 2 teaspoons of 2% lidocaine injection
  Arms: Lidocaine Group
Drug: Placebo — Saline injection
  Arms: Sham Group

SUMMARY:
This research is being done to determine if an anesthetic like Lidocaine, may be effective when injected around the sciatic nerve of the intact limb in patients with limb loss pain on the contralateral side.

ELIGIBILITY:
Inclusion Criteria:

* Lower extremity amputation performed more than 12 months before study enrollment
* PLP/RLP in affected amputated limb > 4 on NRS26
* Pain duration of more than 6 months despite a trial of conservative therapies for at least 2 months, including oral medications, topical medicines, physical therapy, and physical modalities (i.e., heat, cold, transcutaneous electrical nerve stimulation, phonophoresis)
* Willingness to undergo image guided diagnostic nerve block

Exclusion Criteria:

* Refusal / inability to participate or provide consent
* Contraindications to diagnostic nerve block
* Non-neurogenic source of PLP/RLP
* Current opioid use > 50 morphine milligram equivalents per day
* Any interventional pain treatment in the residual limb within the last 30 days
* Severe uncontrolled medical condition (i.e., hypertensive crisis, decompensated hypothyroidism)
* Use of investigational pain drug within past 30 days or other concurrent clinical trial enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in pain | Baseline, 60 minutes post injection
  Measured using self-reported Numerical Rating Scale (NRS) where 0=no pain and 10=worst pain.
Change in Functional Improvement | Baseline, 5 days post-injection
  Measured using self-reported 20-item Orthotic and Prosthetics User's Survey (OPUS) Lower Extremity Functional Status Measurement survey. Total scores range from 0-100 scale with higher scores indicating a better outcome.

SECONDARY OUTCOMES:
Change in disability | Baseline, 5 days post-injection
  Measured using self-reported 18-item The Groningen Activity Restriction Scale (GARS) that is a general disease independent instrument for measuring disability. Total scores range from 18-72. The higher the score the greater the disability.
Change in Pressure-Pain Algometry | Baseline, 5 days post-injection
  Qualified study personnel will measure pain pressure threshold three times at each visit with an algometer on the participant's residual limb at the point of a maximal pain as indicated by the participant during pre-block physical examination, reported in kilopascal (kPa).
Step Count | 5 days post-injection
  Number of daily steps recorded by Modus StepWatch™ or Evolution EvoWalk™ fitted to the participant's prostheses

CONTACTS AND LOCATIONS:
Overall Officials: Cole Cheney, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Health System - Mankato, Mankato, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials